CLINICAL TRIAL: NCT02501980
Title: Searching for Early Detection Biomarkers and to Reduce Mortality Rate of Hepatocellular Cancer (HCC) in Zhongshan City
Brief Title: Hepatocellular Cancer (HCC) Screening in Zhongshan City
Acronym: HCC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Mingfang Ji, Dr. Mingfang Ji, Zhongshan People's Hospital, Guangdong, China
Other Study IDs: HCC-PRO-001
Record Dates: First submitted 2015-06-11; First posted 2015-07-17 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Liver Neoplasms
Keywords: Screening; Hepatocellular Cancer; Biomarker; Mortality rate
MeSH Terms: conditions — Liver Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples

GROUPS / COHORTS (2):
- Screening: All participants will be tested for HBsAg by using serum samples. Among those who are positive for HBsAg, further clinical work-ups including AFP test and ultrasonography for liver exam will be performed. Repeated check-ups will be performed in 6-months among HBsAg positive group and 3-years among HBsAg negative group.
  Interventions: Biological: Biomarker testing and Ultrasonography
- Non-screening: All subjects in this arm will be followed by linkage to Cancer Register and Population Register.

INTERVENTIONS:
Biological: Biomarker testing and Ultrasonography
  Groups: Screening

SUMMARY:
All participants in the selected communities will be tested for HBsAg by using serum samples. Among those who are positive for HBsAg, further clinical work-ups including AFP test and ultrasonography for liver exam will be performed. High risk group will be selected according to the definition. HCC diagnosis will be determined according to imaging and/or biopsy result. Repeated check-ups will be performed in 6-months among HBsAg positive group and 3-years among HBsAg negative group.

All subjects in the control arm (control communities) will be followed by record linkage to Cancer Register and Population Register.

DETAILED DESCRIPTION:
Sample selection

* Select communities of 70,000 to 120,000 populations in Zhongshan City as the investigators' fields.
* Divide them into screening group and control group according to the areas of administration

Participants recruitment

- Subjects voluntarily attend this screening study

Informed consent - Informed consent forms will be collected at the recruitment.

Questionnaires

- Face-to-face interviews are conducted by well-trained investigators

Serological tests

* Each blood samples will be tested for the surface antigen of the hepatitis B virus (HBsAg).
* Among those who are positive for HBsAg, further clinical work-ups including Alpha-Fetoprotein(AFP) test and ultrasonography for liver exam will be performed and high risk group will be selected according to the definition.
* HCC diagnosis will be determined according to imaging and/or biopsy result.
* The rest of the blood samples will be stored at the biobank of Zhongshan People's Hospital.

Follow up

* The cohort will follow up according to the screening protocol. Briefly, Repeated check-ups will be performed in 6-months among HBsAg positive group and 3-years among HBsAg negative group.
* All subjects in the control arm (control communities) will be followed by record linkage to Cancer Register and Population Register.

ELIGIBILITY:
Inclusion Criteria:

* Residences in Zhongshan City
* Have no medical records of hepatocellular cancer
* ECOG 0-2
* Provide written informed consent forms
* Have a good physical and psychological condition

Exclusion Criteria:

* Have severe cardiovascular or kidney disease
* Have medical records of hepatocellular cancer

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy residences in Zhongshan City.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2012-01; Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
5-year HCC specific mortality rate | 10 years
  To reduce 5-year HCC specific mortality rate compare with that of general population

SECONDARY OUTCOMES:
Early diagnosis rate of HCC | 5 years
  To improve early diagnosis rate of HCC compare with that of general population
Identification of early diagnosis markers of HCC | 5 years
  To identify early expression markers of HCC

CONTACTS AND LOCATIONS:
Overall Officials: Mingfang Ji, MD, Principal Investigator — Zhongshan People's Hospital, Guangdong, China
Locations (1):
- Zhongshan People's Hospital, Zhongshan, Guangdong, China